CLINICAL TRIAL: NCT04321772
Title: Effects of Exercise Intensity and Rest Intervals on Intracellular Signals and Anabolic Response of Skeletal Muscle to Resistance Training
Brief Title: Muscle Response to High Intensity Interval Resistance Training (HIIRT)
Acronym: HIIRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova (Other)
Collaborators: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Antonio Paoli, Full Professor, University of Padova
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: HIIRT12
Record Dates: First submitted 2020-03-19; First posted 2020-03-25 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Exercise; Resistance Training
Keywords: resistance training; recovery; muscle hypertrophy; muscle signalling
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Same subjects serve as both the test and control arms which allows for within-subject comparison. Using a within-person design, participants trained each lower limb on separate days under two different training stimulus (HIIRT) and traditional training (TRT)
Who Masked: Outcomes Assessor
Masking Description: The samples analysed were masked by a number without any indication of the arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Intensity Interval Resistance Training (HIIRT) (Experimental): HIIRT technique consisted of three sets of: 6 repetitions at 80% 1RM (1 repetition maximum) and then 20 seconds of rest and 2/3 repetitions (until exhaustion) repeated for 3 times with 2'30" rest between sets; while TRT consisted of 3 sets of 15 reps with 75 sec of rest between sets.
  Interventions: Other: High Intensity Interval Resistance Training
- Traditional Resistance Training (TRT) (Active Comparator): TRT protocol performed 3 series of 15 repetitions at 60% 1RM with 75" of rest between sets.
  Interventions: Other: Traditional Resistance Training

INTERVENTIONS:
Other: High Intensity Interval Resistance Training — Subjects trained one leg with HIIRT
  Arms: High Intensity Interval Resistance Training (HIIRT)
Other: Traditional Resistance Training — Subjects trained the other leg with HIIRT
  Arms: Traditional Resistance Training (TRT)

SUMMARY:
Resistance training (RT) is one of the most important stimuli for muscle hypertrophy and it plays an important role on weight loss and fatty acid oxidation increase. RT affects anabolic pathways but the differences among various training techniques has been till now were poorly investigated. The aim of this study was to compare the effect of two different intensity of training, high-intensity interval resistance training (HIIRT) and traditional resistance training (TRT), on muscle signalling pathway.

DETAILED DESCRIPTION:
Nine young healthy subjects performed HIIRT and TRT protocol in two different moments and with different legs. HIIRT technique consisted of three sets of: 6 repetitions at 6RM (6 repetitions maximum) and then 20 seconds of rest and 2/3 repetitions (until exhaustion) repeated for 3 times with 2'30" rest between sets; while TRT consisted of 3 sets of 15 reps with 75 sec of rest between sets. Biopsies from the vastus lateralis were taken at baseline (pre), immediately (0h) at the end of training, 6 hours (6h) and 24 hours (24h) after training. Western blot and RT-PCR mRNA (Reverse transcriptase-polymerase chain reaction) analysis were performed to assess muscle signalling pathway activation

ELIGIBILITY:
Inclusion Criteria:

* moderate active
* experience with resistance training

Exclusion Criteria:

* history of recent myocardial infarction,
* severe cardiac arrhythmia,
* unstable angina,
* poorly controlled hypertension,
* poorly controlled diabetes mellitus,
* frequent or complex ventricular ectopy which might interfere with one's ability to adhere to exercise protocols

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2012-02-01 (Actual); Primary Completion 2012-05-15 (Actual); Study Completion 2013-02-10 (Actual)

PRIMARY OUTCOMES:
pAMPKThr172 in skeletal muscle tissue measured by immunoblot | 24 hours
  measurement of pAMPKThr172 in skeletal muscle tissue taken by biopsy
pERK 1/2Thr202/Tyr204 in skeletal muscle tissue measured by immunoblot | 24 hours
  measurement of pERK 1/2Thr202/Tyr204 in skeletal muscle tissue taken by biopsy
pS6Ser235/236 in skeletal muscle tissue measured by immunoblot | 24 hours
  measurement of pS6Ser235/236 in skeletal muscle tissue taken by biopsy
p4EBP1Thr37/46 in skeletal muscle tissue measured by immunoblot | 24 hours
  measurement of p4EBP1Thr37/46 in skeletal muscle tissue taken by biopsy
ACC (acetyl-coenzyme A carboxylase) phosphorylation in skeletal muscle tissue measured by immunoblot | 24 hours
  ACC phosphorylation in skeletal muscle tissue taken by biopsy
IGF-1 mRNA (messenger ribonucleic acid) in skeletal muscle tissue measured by Quantitative polymerase chain reaction (qPCR) | 24 hours
  IGF-1 mRNA in skeletal muscle tissue taken by biopsy
IGF-1ea (insulin like growth factor) mRNA in skeletal muscle tissue measured by Quantitative polymerase chain reaction (qPCR) | 24 hoursn
  IGF-1ea mRNA in skeletal muscle tissue taken by biopsy
MGF (mechanical growth factor) mRNA in skeletal muscle tissue measured by Quantitative polymerase chain reaction (qPCR) | 24 hours
  MGF mRNA in skeletal muscle tissue taken by biopsy
STARS mRNA in skeletal muscle tissue measured by Quantitative polymerase chain reaction (qPCR) | 24 hoursn
  STARS mRNA in skeletal muscle tissue taken by biopsy
Myogenin mRNA in skeletal muscle tissue measured by Quantitative polymerase chain reaction (qPCR) | 24 hours
  Myogenin mRNA in skeletal muscle tissue taken by biopsy
IL-6 (interleukin 6) mRNA in skeletal muscle tissue measured by Quantitative polymerase chain reaction (qPCR) | 24 hours
  IL-6 mRNA in skeletal muscle tissue taken by biopsy
PGC1a4 (Peroxisome proliferator-activated receptor gamma coactivator 1-alpha 4) mRNA in skeletal muscle tissue measured by Quantitative polymerase chain reaction (qPCR) | 24 hours
  PGC1a4 mRNA in skeletal muscle tissue taken by biopsy
PGC1a (Peroxisome proliferator-activated receptor gamma coactivator 1-alpha) mRNA in skeletal muscle tissue measured by Quantitative polymerase chain reaction (qPCR) | 24 hours
  PGC1a mRNA in skeletal muscle tissue taken by biopsy
Atrogin mRNA in skeletal muscle tissue measured by Quantitative polymerase chain reaction (qPCR) | 24 hours
  Atrogin mRNA in skeletal muscle tissue taken by biopsy
Beclin mRNA in skeletal muscle tissue measured by Quantitative polymerase chain reaction (qPCR) | 24 hours
  Beclin mRNA in skeletal muscle tissue taken by biopsy
Myostatin mRNA in skeletal muscle tissue measured by Quantitative polymerase chain reaction (qPCR) | 24 hours
  Myostatin mRNA in skeletal muscle tissue taken by biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Paoli, MD, Study Director — University of Padova
Locations (1):
- Nutrition and Exercise Lab, DSB, University of Padova, Padua, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Paoli A. Resistance training: the multifaceted side of exercise. Am J Physiol Endocrinol Metab. 2012 Feb 1;302(3):E387. doi: 10.1152/ajpendo.00541.2011. No abstract available. PMID 22275762
- [Background] Paoli A, Moro T, Marcolin G, Neri M, Bianco A, Palma A, Grimaldi K. High-Intensity Interval Resistance Training (HIRT) influences resting energy expenditure and respiratory ratio in non-dieting individuals. J Transl Med. 2012 Nov 24;10:237. doi: 10.1186/1479-5876-10-237. PMID 23176325
- [Background] Paoli A, Pacelli QF, Cancellara P, Toniolo L, Moro T, Canato M, Miotti D, Reggiani C. Myosin isoforms and contractile properties of single fibers of human Latissimus Dorsi muscle. Biomed Res Int. 2013;2013:249398. doi: 10.1155/2013/249398. Epub 2013 Jul 22. PMID 23971027